CLINICAL TRIAL: NCT06150729
Title: Botulinum A Toxin (OnabotulinumtoxinA) Use in Mexican Pediatric Population With Spasticity Associated With Cerebral Palsy: Phase IV, Observational, Non-Interventional, Prospective, Multicenter Study
Brief Title: Study of Intramuscular Injections of OnabotulinumtoxinA to Assess Change in Disease Activity in Pediatric Participants With Spasticity Associated With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P24-430
Record Dates: First submitted 2023-11-21; First posted 2023-11-29 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Spasticity
Keywords: Spasticity; Cerebral Palsy; OnabotulinumtoxinA
MeSH Terms: conditions — Muscle Spasticity; Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- OnabotulinumtoxinA: Participants will receive OnabotulinumtoxinA as prescribed by their physician.

SUMMARY:
Spasticity is often observed as muscle tightness and stiffness in the upper and/or lower limbs. Upper limb spasticity can interfere with joint movement and its severity can range from mild to severe. This study will assess how effective OnabotulinumtoxinA is in treating pediatric participants with Spasticity. Change in disease activity will be evaluated.

OnabotulinumtoxinA is approved drug for treatment of Spasticity. Approximately 106 pediatric participants aged 2-17 years with spasticity associated with cerebral palsy will be enrolled in approximately 10 sites across Mexico.

Participants will receive OnabotulinumtoxinA as prescribed by their physician in accordance to local label and followed for 12 months.

There is expected to be no additional burden for participants in this trial. Participants will attend regular visits to a hospital or clinic in their routine practice.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral/bilateral, upper/lower limb spasticity associated with cerebral palsy.
* Naïve to OnabotulinumtoxinA treatment and who, according to medical and to the standard clinical practice criteria, will receive OnabotulinumtoxinA.
* Treated only with stable doses of short-acting muscle relaxants can be included in the study, at the investigator's discretion, for at least 30 days prior to treatment starting, under the concept that at the time the steady state of the drug (stable plasma concentrations) will theoretically have been reached.
* Under adjuvant treatment with orthoses and other orthopedic devices can be included in the study.
* Participants with physio/physical therapy can be included.

Exclusion Criteria:

* Previously treated with botulinum toxin for spasticity related to cerebral palsy.
* Diagnosed with Eaton-Lambert syndrome, myasthenia gravis, or other neurological diseases with compromised neuromuscular transmission.
* History of hypersensitivity to the study drug or to any of the excipients in the formulation.
* Evidence of inflammation or infection in the anatomical region selected by the investigator for the study drug administration.
* Participants under treatment with drugs that interfere with neuromuscular transmission which, at the investigator's discretion, contraindicate OnabotulinumtoxinA concomitant administration.
* Have had orthopedic surgery in the segment to be infiltrated in the 12 months prior to drug application.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Participants (2-17 years) with spasticity associated with cerebral palsy.
Sampling Method: Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2025-05-30 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Absolute Total Dose | Up to 12 months
  OnabotulinumtoxinA total dose applied at visit will be assessed.
Total Dose Per Kilogram | Up to 12 months
  OnabotulinumtoxinA total dose applied at each visit, divided by patient's body weight will be assessed.
Dose Per Muscle | Up to 12 months
  OnabotulinumtoxinA dose applied to each muscle, regardless of punctures' number on that muscle will be assessed.
Application Sites Number Per Muscle | Up to 12 months
  Number of puncture sites per muscle will be assessed.
Re-administration Interval | Up to 12 months
  Re-administration interval is defined as number of days between drug application and previous application.
Needle Gauge | Up to 12 months
  Needle gauge is defined as diameter of needle thickness with which study treatment is applied.
Needle Length | Up to 12 months
  Needle length is defined as distance from the needle base to the needle bevel tip.
Preventive Pain Management Technique | Up to 12 months
  Type of method used to control procedural pain will be assessed.
Method to Locate Application Site | Up to 12 months
  Type of method used to identify muscle and treatment application site will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (8):
- Mexico (8):
  - Hospital General Regional 180 IMSS /ID# 261458, Guadalajara, Jalisco
  - Clinica de Rehabilitacion Integral Yupi /Id# 261461, Puerto Vallarta, Jalisco
  - Hospital General ISSSTE Tacuba /ID# 261460, Mexico City, Mexico City
  - Hospital General ISSSTE Tacuba /ID# 261932, Mexico City, Mexico City
  - Cree Dif Nuevo Leon /Id# 261454, Monterrey, Nuevo LEON, Nuevo León
  - Hospital Militar De Zona De Villahermosa /ID# 261451, Villahermosa, Tabasco
  - Cri Dif Jalisco /Id# 261459, Guadalajara
  - Crit Estado de México /Id# 261934, Tlalnepantla

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=P24-430